CLINICAL TRIAL: NCT05187884
Title: Neoadjuvant/Adjuvant Trial of Darovasertib in Ocular Melanoma
Acronym: NADOM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Anthony Joshua, FRACP, Head of Medical Oncology, St Vincent's Hospital, Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NADOM
Record Dates: First submitted 2021-12-09; First posted 2022-01-12 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Ocular Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Darovasertib 300mg bd
  Interventions: Drug: Darovasertib

INTERVENTIONS:
Drug: Darovasertib — Oral Darovasertib 300 mg tablets twice daily

SUMMARY:
The purpose of this study is to determine the feasibility and tolerability of neo-adjuvant/adjuvant Darovasertib on uveal melanoma patients.

Who is it for? Patients may be eligible to join this study with high-risk uveal melanoma and planned to undergo enucleation

Study details:

Eligible patients will undergo up to 4 weeks of treatment with Darovasertib (300mg, twice a day as a starting dose) and once determiend safe then up to 6 months after fulfilling inclusion/exclusion criteria and consent. Select patients will undergo adjuvant treatment for 6 months based on their initial response.

It is hoped that this research will provide insight into the safety and tolerability of Darovasertib. Furthermore, it aims to document the pharmacodynamic and pharmacokinectic effects of Darovasertib on uveal melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age.
* Primary diagnosis of uveal melanoma as clinically determined by the treating investigator planned for enucleation (prior plaque brachytherapy is permitted)
* Patient is able to provide written, informed consent before initiation of any study related-procedures, and is able, in the opinion of the investigator, to comply with all the requirements of the study.
* Life expectancy > 3 months.
* Able to safely swallow orally administered medication.
* Patients with a prior history of or clinically stable concurrent malignancy are eligible for enrolment provided the malignancy is clinically insignificant, no treatment is required, and the patient is clinically stable

  * Patients with a history of squamous or basal cell carcinoma of the skin or carcinoma in the situ of the cervix may be enrolled.
  * Patients with prostate cancer with an elevated PSA not requiring treatment may be enrolled
* Patient has Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1 (Karnofsky = 70%).
* Patient has adequate organ function at screening:

  * Absolute neutrophil count = 1500/mm3 without the use of hematopoietic growth factors
  * Platelet count = 75,000/mm3 (must be at least 2 weeks post-platelet transfusion and not receiving platelet-stimulating agents)
  * Haemoglobin = 8.0 g/dL (must be at least 2 weeks post-red blood cell transfusion and not receiving erythropoietic-stimulating agents)
  * Total bilirubin = 1.5 x the upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) = 3 x ULN in the absence of documented liver metastases
  * Serum albumin = 30 umol/L
  * Creatinine Clearance = 60 mL/min/1.73 m2 by Cockroft-Gault equation [Appendix 6]
  * Prothrombin time/International Normalized Ratio (INR) or partial thromboplastin time test results at screening = 1.5 x ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose for at least 4 weeks prior to the first dose of study drug).
* Female patients of childbearing potential must be non-pregnant, non-lactating, and have a negative serum human chorionic gonadotropin pregnancy test result within 28 days prior to the first study drug administration.

  * Females of childbearing potential who are sexually active with a non-sterilized male partner agree to use effective methods of contraception from screening, throughout the study drug and agree to continue using such precautions for 30 days after the final dose of study drug.
  * Non-sterilized males who are sexually active with a female of childbearing potential must agree to use effective methods of contraception from Day 1 throughout the study drug and for 30 days after the final dose of study drug.

Exclusion Criteria:

* Previous treatment with a PKC inhibitor
* Have AEs from prior anti-cancer therapy that have not resolved to Grade =1 except for alopecia, prior peripheral neuropathy, or anaemia. Endocrinopathies resulting from previous immunotherapy are considered part of the medical history and not an AE.
* Untreated or symptomatic malignant lesions in the central nervous system (CNS).
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) - related illness.
* Active infection requiring therapy (except nail fungus), positive tests for Hepatitis B surface antigen (HBsAg) with detected Hepatitis B virus (HBV) DNA or positive Hepatitis C antibody with detected Hepatitis C virus (HCV) RNA.
* Prior gastrectomy or upper bowel removal or any other gastrointestinal disorder or defect e.g., malabsorption disorder such as Crohn's disease or ulcerative colitis, that would interfere with absorption of Darovasertib.
* Patients who are receiving treatment with medications that cannot be discontinued prior to study entry and that are considered to be any of the following (see Appendix 4):

  * known to be strong inducers or inhibitors of CYP3A4/5
  * known to be substrates of CYP3A4/5, OAT3, OATP1B1, and MATE1/2-Kwith a narrow therapeutic index
* Females who are pregnant or breastfeeding:

  * Women of childbearing potential must not be considering getting pregnant during the study.
  * Patients of reproductive potential (male & female) must practice an effective method of contraception during treatment and for 30 days following the last dose of Darovasertib. Patients unwilling to do so will be excluded.
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * History or presence of ventricular tachyarrhythmia
  * Presence of unstable atrial fibrillation (ventricular response > 100 BPM); patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria
  * Angina pectoris or acute myocardial infarction = 6 months prior to starting study drug
  * Other clinically significant heart disease (e.g., symptomatic congestive heart failure; uncontrolled arrhythmia or hypertension; history of labile hypertension or poor compliance with an antihypertensive regimen)
  * Patients with a drug eluting stent for cardiovascular purposes placed = 6 months prior to starting study drug
  * Corrected QT interval using Fridericia's method (QTcF) > 480 msec on baseline ECG (mean of baseline values). If electrolytes are abnormal, they may be corrected, and baseline ECGs should be repeated (Appendix 5).
* Known to have previously received Darovasertib
* Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the opinion of the investigator, would make the patient inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of a up to a 56-day course of Darovasertib via clinical assessment by CTCAE v5.0 guidelines for adverse event(s) | 56 days post commencement of investigational product.
  Safety Profile
Percentage of participants that complete the 56-day treatment period. | 56 days post commencement of investigational product.

SECONDARY OUTCOMES:
To determine the effect of neo-adjuvant Darovasertib on tumour size in uveal melanoma as measured by ocular ultrasound. | 56 days
To explore time to recurrence/disease-specific survival in patients on adjuvant Darovasertib assessed by standard of care imaging measured using RECIST 1.1. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, FRACP, MBBS, PhD, Principal Investigator — St Vincent's Hospital, Sydney
Locations (2):
- Australia (2):
  - Kinghorn Cancer Centre, St. Vincent's Hospital, Sydney, New South Wales
  - Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
No Plan to share participant data with individuals outside this trial